CLINICAL TRIAL: NCT04125810
Title: A Randomized, Triple-blind, Placebo-controlled, Parallel-groups Clinical Trial to Assess the Safety and Efficacy of Lactobacillus Paracasei (Lpc-37) to Modulate Psychological Stress
Brief Title: A Study to Assess the Safety and Efficacy of Probiotic to Modulate Psychological Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: ICON plc (Industry); Daacro (Network); 4Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NH03821
Record Dates: First submitted 2019-08-30; First posted 2019-10-14 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Stress, Psychological; Healthy
Keywords: Probiotic; Stress; Gut-brain axis
MeSH Terms: conditions — Stress, Psychological | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Probiotic
  Interventions: Biological: Probiotic
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Probiotic — Probiotic
  Arms: Probiotic
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to determine whether Probiotic can modulate the psychological stress experienced by healthy medical, dental and health science students preparing for university/institute of technology semester examination (s), measured by self-report scales and hypothalamic pituitary adrenal axis activity, compared with placebo.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to determine whether Probiotic can modulate the psychological stress experienced by healthy medical, dental and health science students preparing for university/institute of technology semester examination (s), measured by self-report scales and hypothalamic pituitary adrenal axis activity, compared with placebo.

The target group of the proposed study will consist of stress vulnerable / sensitive, healthy male and female adult participants currently enrolled in medical, dental or health science university course that are experiencing psychological stress induced by preparation for university/institute of technology semester examination (s).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, informed consent to participate in the study
2. Currently enrolled in medical, dental or health science university/institute of technology course with intention to sit semester examination(s)
3. Male or female aged between 18-40 years (inclusive)
4. Body mass index (BMI) between 18.5 - 29.9 Kg/m2
5. Blood, urine and gastrointestinal safety parameters and blood pressure measurement at baseline indicate they are healthy in the opinion of the Principal Investigator
6. In good general health as estimated by the Principal Investigator, based on medical history (self-reported)
7. Ability of the participant (in the Principal Investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
8. Ability of the participant (in the Principal Investigator's opinion) to fully comprehend and self-complete all participant reported outcomes (in UK English language)
9. Participant is willing to maintain habitual diet (including caffeine and alcohol), physical activity patterns and smoking habits throughout the intervention period
10. Agreement to comply with the protocol and study restrictions
11. Available for all study visits
12. Females of child-bearing potential required to provide a negative urine pregnancy test and be using effective contraception (e.g. surgically sterilized (tubal ligation or hysterectomy or partner is post-vasectomy, with sterility confirmed) or use an intrauterine device (IUD), a diaphragm or condom combined with contraceptive sponge, foam or jelly, or be using an oral contraceptive for at least 2 cycles before the screening visit (Visit 2). Women who are in same sex relationships or abstaining from sex are not required to take a pregnancy test or be using effective contraception
13. Male participants must agree to use a condom during sexual intercourse from Visit 3 onwards
14. Covered by health insurance system and / or in compliance with the recommendations of National Law in force relating to biomedical research

Exclusion Criteria:

1. Suspected diagnosis of one or more DSM-IV axis 1 disorder(s), including but not limited to: current major depression, anxiety disorder, bipolar spectrum disorder or schizophrenia, as determined by MINI International Neuropsychiatric Interview (MINI) and/or currently diagnosed with one or more DSM-IV axis 1 disorder(s), per Diagnostic and Statistical Manual of Mental Disorders, 4th Edition.
2. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal (irritable bowel syndrome (IBS), inflammatory bowel disease (IBD)), immunological, metabolic (including diabetes and cardiovascular disease), neurodevelopmental or any condition which contraindicates, in the Principal Investigator's judgement, entry to the study
3. Currently taking (from Visit 1 onwards) or have previously taken (last 4 weeks prior to Visit 1) psychoactive medication (anxiolytics, sedatives, hypnotics, anti-psychotics, anti-depressants, anti-convulsants, centrally acting corticosteroids, opioid pain relievers)
4. Currently taking (from Visit 1 onwards) medication or dietary supplements that the Principal Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results (e.g. melatonin, St. John's Wort, Rescue® products including Rescue Remedy®, Rescue® Energy, Rescue® Pastilles, Rescue® Pearls, Rescue Sleep® Rescue PlusTM, omega-3 dietary supplements (including fish oil), Cannabidiol (CBD), non-steroidal anti-inflammatory drugs (NSAIDS), over-the-counter sleep medication (not categorized as sedatives, hypnotics or anti-depressants), anti-coagulants, anti-cholinergic drugs or acetylcholinesterase inhibitors, proton pump inhibitors, anti-histamines that cause drowsiness, pseudoephedrine)
5. Recent (within last 4 weeks prior to Visit 1) or ongoing antibiotic therapy
6. Currently taking (from Visit 1 onwards) concentrated sources of probiotics and/or prebiotics other than the provided study products (e.g., probiotic/prebiotic tablets, capsules, drops or powders), including yoghurt / yoghurt drinks
7. Pregnant or lactating female, or pregnancy planned during the intervention period
8. Have self-reported dyslexia
9. History of or current alcohol, drug, or medication abuse (self-reported)
10. Self-declared illicit drug users (including cannabis and cocaine) in the past 1 month prior to Visit 1
11. Excessive alcohol consumption (consuming > 8 units of alcohol for men and > 6 units of alcohol for women in a single session) > 3 times per week for 3 weeks prior to Visit 1
12. Significant change in tobacco, snuff, nicotine or e-cigarette usage habits in the past 1 month before Visit 1 or planned cessation of the use of these products during the intervention period
13. Contraindication to any substance in the investigational product
14. Participation in another study with any investigational product or drug within 60 days of Visit 1
15. Principal Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study
16. Participant under administrative or legal supervision
17. Previous participation in the ChillEx study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory (STAI)-state total score | from baseline to 8 weeks
  Absolute change in STAI-state total score between the active versus placebo group

SECONDARY OUTCOMES:
Change in Cortisol awakening response (CAR) | from baseline to 8 weeks
  The absolute changes in the CAR will be analyzed in the same fashion as described for the primary variable.
Change in perceived stress (Visual Analog Scale (VAS)-stress) | from baseline to 8 weeks
  The absolute change in VAS-stress score will be analyzed in the same fashion as described for the primary variable.
  * Visual Analog Scale (VAS)-stress.
  * Participants indicate on a 100mm line how stressed they perceived themselves to be over the last week. The scale is anchored from 0 = felt not stressed at all to 100 = felt highly stressed. Scores are determined by measuring from the left end to the mark using a ruler.
Change in DASS-21, depression scale score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in DASS-21, depression scale score will be analyzed in the same fashion as described for the primary variable.
  * Depression, anxiety, stress scale (21 items).
  * The DASS gives information about negative emotional states of depression, anxiety and stress. The questionnaire includes 3 scales (depression, anxiety and stress) of which each scale includes 7 items that are divided into subscales of 2-5 items of similar content.
Change in DASS-21, anxiety scale score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in DASS-21, anxiety scale score will be analyzed in the same fashion as described for the primary variable.
  * Depression, anxiety, stress scale (21 items).
  * The DASS gives information about negative emotional states of depression, anxiety and stress. The questionnaire includes 3 scales (depression, anxiety and stress) of which each scale includes 7 items that are divided into subscales of 2-5 items of similar content.
Change in DASS-21, stress scale score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in DASS-21, stress scale score will be analyzed in the same fashion as described for the primary variable.
  * Depression, anxiety, stress scale (21 items).
  * The DASS gives information about negative emotional states of depression, anxiety and stress. The questionnaire includes 3 scales (depression, anxiety and stress) of which each scale includes 7 items that are divided into subscales of 2-5 items of similar content.
Change in HADS, depression score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in HADS, depression score will be analyzed in the same fashion as described for the primary variable.
  * Hospital anxiety and depression scale.
  * The HADS is a 14 item self-report screening tool which is widely used in the clinic to assess levels of depression and anxiety.
Change in HADS, anxiety score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in HADS, anxiety score will be analyzed in the same fashion as described for the primary variable.
  * Hospital anxiety and depression scale.
  * The HADS is a 14 item self-report screening tool which is widely used in the clinic to assess levels of depression and anxiety.
Change in PSS, total score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in PSS, total score will be analyzed in the same fashion as described for the primary variable.
  * Cohen's perceived stress scale.
  * The PSS is a self-report measure in which participants rate, on a 5-point scale ranging from 0 (never) to 4 (very often), how often they have particular thoughts or feelings described by each of the 10 items.
  * Scores range from 0-40, with higher scores indicating greater stress over the previous month.
Change in BL-VAS, alertness score from baseline (Visit 3) to 8 weeks (Visit 5) | from baseline to 8 weeks
  The absolute changes in BL-VAS, alertness score will be analyzed in the same fashion as described for the primary variable.
  * Bond-Lader visual analogue scale.
  * The Bond-Lader VAS consist of 16 scales with anchors of related mood/ arousal dimensions (e.g. calm-excited; strong-feeble).
  * Participants indicate on a 100mm line how they feel along each mood dimension at that specific time, and scores from the 16 scales are converted into three composite mood/ arousal dimensions; alertness, calmness and contentedness.
Change in BL-VAS, contentment score | from baseline to 8 weeks
  The absolute changes in BL-VAS, contentment score will be analyzed in the same fashion as described for the primary variable.
Change in BL-VAS, calmness score | from baseline to 8 weeks
  The absolute changes in BL-VAS, calmness score will be analyzed in the same fashion as described for the primary variable.
Change in Pittsburgh Sleep Quality Index (PSQI), total score | from baseline to 8 weeks
  The absolute changes in the PSQI, total score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, duration of sleep score | from baseline to 8 weeks
  The absolute changes in the PSQI, duration of sleep score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, sleep disturbance score | from baseline to 8 weeks
  The absolute changes in the PSQI, sleep disturbance score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, sleep latency score | from baseline to 8 weeks
  The absolute changes in the PSQI, sleep latency score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, daytime dysfunction due to sleepiness score | from baseline to 8 weeks
  The absolute changes in the PSQI, daytime dysfunction due to sleepiness score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, sleep efficiency score | from baseline to 8 weeks
  The absolute changes in the PSQI, sleep efficiency score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, subjective sleep quality score | from baseline to 8 weeks
  The absolute changes in the PSQI, subjective sleep quality score will be analyzed in the same fashion as described for the primary variable.
Change in PSQI, use of medication sleep score | from baseline to 8 weeks
  The absolute changes in the PSQI, use of medication sleep score will be analyzed in the same fashion as described for the primary variable.
Change in evening cortisol | from baseline to 8 weeks
  Evening cortisol: Participants will provide x1 saliva sample each evening during two consecutive working days at approximately 8pm prior to Visit 3, Visit 4, Visit 5 and Visit 6.
  Concentrations of cortisol will be assayed in saliva supernatants using ELISA kits specifically designed for cortisol quantification, following manufacturer's instructions.

OTHER OUTCOMES:
IPAQ-short, physical activity level score | from baseline to 4 weeks, 8 weeks and 10 weeks
  Changes in International Physical Activity Questionnaire (IPAQ)-short, physical activity level score
Detection of Probiotic in feces | from baseline to 8 weeks
  Changes in detection of Probiotic in feces
STAI-state | from baseline to 4 weeks and 10 weeks
  Changes in State-trait anxiety inventory (STAI)-state, total score
Changes in Cortisol awakening response (CAR) | from baseline to 4 weeks and 10 weeks
  Cortisol awakening response: Participants will provide x3 saliva samples each morning during two consecutive working days prior to Visit 3, Visit 4, Visit 5 and Visit 6.
  Concentrations of cortisol will be assayed in saliva supernatants using ELISA kits specifically designed for cortisol quantification, following manufacturer's instructions.
Changes in evening cortisol | from baseline to 4 weeks and 10 weeks
  Evening cortisol: Participants will provide x1 saliva sample each evening during two consecutive working days at approximately 8pm prior to Visit 3, Visit 4, Visit 5 and Visit 6.
  Concentrations of cortisol will be assayed in saliva supernatants using ELISA kits specifically designed for cortisol quantification, following manufacturer's instructions.
Changes in Visual Analog Scale (VAS)-stress (VAS-stress) | from baseline to 4 weeks and 10 weeks
  Visual Analog Scale (VAS)-stress (VAS-stress): Participants will complete the VAS-stress at clinic visits 2, 3, 4, 5 and 6. Participants indicate on a 100mm line how stressed they perceived themselves to be over the last week. The scale is anchored from 0 = felt not stressed at all to 100 = felt highly stressed. Scores are determined by measuring from the left end to the mark using a ruler.
Depression, anxiety, stress scale (21 items) (DASS-21) | from baseline to 4 weeks and 10 weeks
  * DASS-21, depression scale score
  * DASS-21, anxiety scale score
  * DASS-21, stress scale score
  Participants will complete the DASS-21 at clinic visits 2, 3, 4, 5 and 6. The DASS gives information about negative emotional states of depression, anxiety and stress. The questionnaire includes 3 scales (depression, anxiety and stress) of which each scale includes 7 items that are divided into subscales of 2-5 items of similar content.
Hospital anxiety and depression scale (HADS) | from baseline to 4 weeks and 10 weeks
  * HADS, depression score
  * HADS, anxiety score
  Participants will complete the HADS at clinic visit 2, 3, 4, 5 and 6. The HADS is a 14 item self-report screening tool which is widely used in the clinic to assess levels of depression and anxiety. It was developed as a tool for quick and easy use in a hospital setting, but has since been validated in primary care and in the community.
Cohen's perceived stress scale (PSS) | from baseline to 4 weeks and 10 weeks
  o PSS, total score
  Participants will complete the PSS at clinic visits 2, 3, 4, 5 and 6. The PSS is a self-report measure in which participants rate, on a 5-point scale ranging from 0 (never) to 4 (very often), how often they have particular thoughts or feelings described by each of the 10 items. Scores range from 0-40, with higher scores indicating greater stress over the previous month.
Bond-Lader visual analogue scale (BL-VAS) | from baseline to 4 weeks and 10 weeks
  * BL-VAS, alertness score
  * BL-VAS, contentment score
  * BL-VAS, calmness score
  Participants will complete the BL-VAS at clinic visits 2, 3, 4, 5 and 6. The Bond-Lader VAS consist of 16 scales with anchors of related mood/ arousal dimensions (e.g. calm-excited; strong-feeble). Participants indicate on a 100mm line how they feel along each mood dimension at that specific time, and scores from the 16 scales are converted into three composite mood/ arousal dimensions; alertness, calmness and contentedness.
Pittsburgh sleep quality index (PSQI) | from baseline to 4 weeks and 10 weeks
  * PSQI, total score; PSQI, duration of sleep score
  * PSQI, sleep disturbance score
  * PSQI, sleep latency score
  * PSQI, daytime dysfunction due to sleepiness score
  * PSQI, sleep efficiency score
  * PSQI, subjective sleep quality score
  * PSQI, use of medication sleep score
  Participants will complete the PSQI at clinic visits 2, 3, 4, 5 and 6. The PSQI assesses sleep quality over the prior month. It is a self-report measure comprised of 19 items which are designed to measure 7 key components indicating either problematic or non-problematic sleep; sleep latency, sleep duration, sleep efficiency, sleep disturbances, subjective sleep quality, use of sleep medication and daytime dysfunction due to sleep disturbance. Scores on each component are combined to give a global score. Scores ≥5 indicate significant disturbances of sleep during the prior month.
Fecal microbiota composition | from baseline to 8 weeks
  Changes in fecal microbiota composition
Compliance of study product | 10 weeks
  Compliance of study product
  * Participants will be asked to return the remaining study products to the study site at each visit during the intervention period (Visit 4, 5 and 6) for study product accountability and accurate determination of compliance throughout the intervention period.
  * A study product inventory (dispensing records) will be used by site staff to record all study product dispensed and returned.

CONTACTS AND LOCATIONS:
Overall Officials: Balgit Chhokar, Study Director — Medinova East London Dedicated Research Center
Locations (7):
- Atlantia Food Clinical Trials Ltd, Cork, Ireland
- United Kingdom (6):
  - MediNova Warwickshire Dedicated Research Centre, Kenilworth
  - MediNova North London Dedicated Research Centre, Northwood
  - MediNova Research East London Clinical Studies Centre, Romford
  - MediNova Yorkshire Dedicated Research Centre, Shipley
  - MediNova South London Dedicated Research Centre, Queen Mary's Hospital, Sidcup
  - MediNova West London Dedicated Research Centre, Wokingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Makela SM, Griffin SM, Reimari J, Evans KC, Hibberd AA, Yeung N, Ibarra A, Junnila J, Turunen J, Beboso R, Chhokar B, Dinan TG, Cryan J, Patterson E. Efficacy and safety of Lacticaseibacillus paracasei Lpc-37(R) in students facing examination stress: A randomized, triple-blind, placebo-controlled clinical trial (the ChillEx study). Brain Behav Immun Health. 2023 Aug 1;32:100673. doi: 10.1016/j.bbih.2023.100673. eCollection 2023 Oct. PMID 37662485